CLINICAL TRIAL: NCT03900702
Title: Training Foundational Skills to Enhance Cognition in Older Adults
Brief Title: Training to Enhance Cognition in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeanne Townsend, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Jeanne Townsend, PhD, Professor Emeritus, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U01AG062371 (NIH); U01AG062371 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Cognitive Enhancement; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Active Comparator): Gaze-driven games, played at home on PC with eye-tracker, to train resistance to attention distraction and speed of processing.
  Interventions: Behavioral: Gaze-driven training games
- Wait List Control (No Intervention): Wait list then cross over to active intervention.

INTERVENTIONS:
Behavioral: Gaze-driven training games — Training games are played on a PC with attached eye-tracker. Games include embedded training principles to improve attentional control including resistance to distraction and inhibitory control.
  Arms: Active Intervention

SUMMARY:
This is a planning project with a clinical trial pilot to prepare for a larger fully powered clinical trial. Goals of this pilot project are: to identify and address any modifications of the games required for adaptation to diminished sensory abilities; to optimize training dosage and test timing of retention of effects; and to test and refine the battery of outcome assessments. Primary outcome assessment are tests of attention distraction (subtest from a Useful Field of View Test). This pilot will explore a number of secondary outcome measures including EEG and functional imaging biomarkers of change, measures of general cognitive improvement and measures of function including a driving simulator task.

DETAILED DESCRIPTION:
This is a planning trial to optimize procedures for a larger clinical trial. Participants will be randomized into one of two groups--an active group that has intervention training after initial visit and a wait control group that begins intervention after 12 weeks. All participants will receive in-lab baseline testing including IQ (WASI-II), a medical/psychiatric history questionnaire, a depression screen (Geriatric Depression Scale Short Form) and a pre-training battery that includes selected tests from the NIH toolbox, the Repeatable Battery for Neuropsychological Status (RBANS), a Useful Field of View task (UFOV), a driving simulator task, a dual (motor-cognitive) task, an n-back task with and without distractors(with EEG) and 6 minutes of resting state EEG. Participants will be trained to use the game system and play the game at the pre-training in-lab visit. Participants will be provided with a PC with eye-tracker that has training game software installed. Participants will play intervention training games at home for 8-12 weeks with in-lab assessments (the pre-training battery described above). Participants will be asked to play the training games a minimum of 5 times per week for 30 minutes at a time. Compliance will be monitored daily over a secure internet connection. If a participant has played less than the required time in a given week, a research associate will contact the participant to inquire about potential problems and to encourage the participant to resume or increase training time. The first group of 36 participants will receive post-training assessments at 8 weeks, 12 weeks and 6 months. The second group of 36 participants will have an additional pre-training session with structural and functional imaging and will receive only pre- and post-training assessment.

ELIGIBILITY:
Inclusion Criteria:

1. age 60-80 years old
2. not demented
3. living independently; and (4) fluent in English.

Exclusion Criteria:

1. history of dementia, stroke, head injury involving loss of consciousness
2. current psychiatric or neurological disorders other than depression/anxiety

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
UFOV Attention Distraction | 12 weeks
  Subtest from Useful Field of View Task
UFOV Speed of Processing | 12 weeks
  Subtest from Useful Field of View Task

SECONDARY OUTCOMES:
Repeatable Battery for Neuropsychological Status (RBANS) | 12 weeks
  Battery to assess general cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Townsend, PhD, Principal Investigator — UCSD
Locations (1):
- Research on Autism and Development Lab, UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available by request to the PI 1 year following completion of study. Materials generated under the project will be disseminated in accordance with University/Participating institutional and NIH policies. Depending on such policies, materials may be transferred to others under the terms of a material transfer agreement. Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data available 1 year following study completion and for 5 years subsequently.
Access Criteria: Access for research or educational purposes, by application specifying use.